CLINICAL TRIAL: NCT03772730
Title: A Multi-Center, Prospective Observational Study to Evaluate the Use of Patient-Specific Precision Injury Signatures to Optimize Orthopaedic Interventions in Multiply Injured Patients
Brief Title: Patient-Specific Precision Injury Signatures in Multiply Injured Orthopaedic Patients
Acronym: PRECISE
Status: Completed | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 00008259
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pelvic, Acetabular, Femur, or Diaphyseal Tibial Operative Orthopaedic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Multiply injured patients having at least one operative orthopaedic injury to the pelvis, acetabulum, femur, or diaphyseal tibia with planned definitive fixation to occur prior to discharge.

SUMMARY:
The purpose of this study is to evaluate the use of precision methods that quantify injury and response to injury to predict how short-term clinical outcomes are affected by initial and staged orthopaedic interventions in multiply injured patients (MIPs) who sustain major orthopaedic trauma.

DETAILED DESCRIPTION:
There is currently a knowledge gap regarding in the treatment of the severely injured MIP, as clinicians are often challenged by when non-life threatening orthopaedic procedures should be performed. Information to guide orthopaedic interventions in MIPs is based primarily on resuscitation parameters and injury severity metrics.Lack of consensus among surgeons regarding choices of orthopaedic interventions reflects the paucity of data to form treatment decisions.

This study will define the key parameters affecting these decisions in a quantitative manner by exploring the efficacy of a precision medicine approach to guide surgical decisions in multiply injured patients (MIPs) with skeletal trauma. According to the National Institutes of Health (NIH),36 precision medicine is "an emerging approach for disease treatment and prevention that takes into account individual variability in genes, environment, and lifestyle for each person." This approach will allow clinicians and researchers to predict more accurately which treatment and prevention strategies for a particular disease will work in which groups of people. The application of precision medicine will bring to bear evidence-based tools that can guide decisions facing the treating surgeons regarding the optimal timing of definitive fracture surgery after injury, as well as defining the magnitude of surgical intervention which may be pursued without engendering clinical complications.

Specific Aim 1: Define groups of patients based on Precision Injury Signatures (mechanical and ischemic injury characteristics and immunologic response profile) that correspond to the following short term clinical outcomes;

1. Multiple organ dysfunction
2. Nosocomial infection
3. Wound complications
4. Resource utilization (ICU/hospital LOS, days on mechanical ventilation, discharge disposition)
5. Death

Hypothesis 1: Patients who develop complicated short term outcomes will demonstrate distinct Precision Injury Signatures compared to patients who have uncomplicated outcomes for injuries of similar magnitude.

Specific Aim 2: Evaluate the impact of timing and magnitude of orthopaedic surgical interventions on progression of patient-specific physiologic and immunologic response. Describe changes in physiologic and immunologic response after initial and staged orthopaedic interventions.

Hypothesis 2: Immunologic and physiologic response to surgery will be a function of initial Precision Injury Signature and timing/magnitude of orthopaedic surgical interventions.

Specific Aim 3: To develop surgical decision rules related to timing of definitive orthopaedic intervention that optimize short term clinical outcomes.

Hypothesis 3a: Initial Precision Injury Signatures can be used to identify orthopaedic trauma patients who are best treated with early definitive treatment or staged definitive intervention.

Hypothesis 3b: Progression of Precision Injury Signatures can be used to determine optimal timing and choices of definitive orthopaedic interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ages 18 years old to 55 years old inclusive;
2. Direct admission to hospital from scene of injury, or if transferred, admitted no more than 6 hours from injury
3. Full trauma activation with either direct admission to Intensive Care Unit (ICU) or other higher level of care, or taken directly to surgery and admitted to ICU after surgery;
4. Sustaining at least one operative orthopaedic injury to the pelvis, acetabulum, femur, or diaphyseal tibia with planned definitive fixation to occur prior to discharge.

Exclusion Criteria:

1. Non-survivable head trauma.
2. Signs of severe traumatic brain injury indicated by a GCS of < 7 at the time of admission and no improvement in the GCS by the time of consent.
3. Spinal cord injury with likely permanent neurologic deficits
4. Pre-existing organ dysfunction or failure prior to their injury, including but not limited to end-stage renal disease, liver failure, congestive heart failure, or severe COPD requiring home oxygen.
5. Qualifying orthopaedic injury primarily a periarticular fracture (tibial pilon or plateau) with planned delay to definitive fixation for soft tissue reasons.
6. Primary blood draw could not be obtained within 3 hours of presentation
7. Patient is pregnant
8. Patient is a prisoner/incarcerated
9. Patient or legally authorized representative (LAR) unable to provide consent prior to 48 hour blood draw.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult (18-55) patients sustaining multiple injuries, including at least one qualifying orthopaedic injury to the pelvis, acetabulum, femur, or diaphyseal tibia.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes recorded during 6month post injury medical record review | 6 months post injury
  Number of occurrences of multiple organ dysfunction, nosocomial infection, wound complications, resource utilization and death as noted in medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Todd McKinley, MD, Principal Investigator — Indiana University/Methodist Hospital
Locations (8):
- United States (8):
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Methodist Hospital/Indiana University, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Carolinas Medical Center, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Health: The University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - University of Washington Harborview Medical Center, Seattle, Washington